CLINICAL TRIAL: NCT03410160
Title: Predisposing Factors for the Incidence of Adrenal Crisis in Chronic Adrenal Insufficiency
Brief Title: Predisposing Factors for the Incidence of Adrenal Crisis
Acronym: PIA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PIA
Record Dates: First submitted 2018-01-18; First posted 2018-01-25 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Adrenal Insufficiency
Keywords: adrenal crisis; predisposing factors
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Retention of samples with and without DNA (whole-blood and serum).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High frequency of adrenal crisis: Patients with a high frequency of adrenal crisis in the past. Intervention: Clinical and biochemical examination (physical examination and blood-sampling before and after oral ingestion of glucocorticoids).
  Interventions: Diagnostic Test: Clinical and biochemical examination.
- Low frequency of adrenal crisis: Patients with no adrenal crisis or a low frequency of AC in the past. Intervention: Clinical and biochemical examination (physical examination and blood-sampling before and after oral ingestion of glucocorticoids).
  Interventions: Diagnostic Test: Clinical and biochemical examination.

INTERVENTIONS:
Diagnostic Test: Clinical and biochemical examination. — Patients with chronic adrenal insufficiency were assessed by clinical and biochemical examination as well as questionnaire to evaluate the quality of hormone replacement therapy with glucocorticoids, education status, cortisol-metabolism, catecholamine deficit, chronic inflammation and variations of the glucocorticoid receptor.

SUMMARY:
Within this clinical study patients with chronic adrenal insufficiency will be investigated by clinical and biochemical examination as well as questionnaire to identify predisposing factors for adrenal crisis.

DETAILED DESCRIPTION:
Patients with chronic adrenal insufficiency (AI) are at risk of suffering from life-threatening adrenal crisis (AC), despite established hormone replacement therapies and patient education. Recent retrospective analyses observed different risk factors for AC, e.g. primary AI and comorbidities. Furthermore, patients that already experienced an AC seem to have an increased risk to develop further AC. The aim of the study is to evaluate potential risk factors/predisposing factors for AC in patients with chronic primary and secondary AI (PAI/SAI). Patients with chronic AI are assessed by clinical and biochemical examination and questionnaire to evaluate the quality of hormone replacement therapy with glucocorticoids, education status, cortisol-metabolism, catecholamine deficit, chronic inflammation and variations of the glucocorticoid receptor. AI patients with a high frequency of AC will be compared to matched controls (age, sex and cause of AI) with no AC or a low frequency of AC in the past.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patient´s written informed consent
* Ability to comply with the protocol procedures
* Patients with chronic primary or secondary adrenal insufficiency under established stable replacement therapy (disease duration at least 2 years)

Exclusion Criteria:

* Age <18 years
* Pregnancy or breast feeding
* Intake of CYP3A4-inducting-drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic adrenal insufficiency under hormone replacement therapy with glucocorticoids.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Chronic inflammation (hsCRP, Interleukin-6) | 1 day
  Measurement of hsCRP (mg/dl) and Interleukin-6 (pg/ml) levels. Hypothesis: Patients with chronic adrenal insufficiency and a high frequency of adrenal crisis exhibit higher hsCRP and Interleukin-6 levels.
Cortisol metabolism | 1 day
  Measurement of cortisol-levels (mg/dl) before as well as 60 min and 120 min after ingestion of hydrocortisone. Hypothesis: Patients with chronic adrenal insufficiency and a high frequency of adrenal crisis exhibit a faster hydrocortisone metabolism.
Replacement therapy with glucocorticoids | 1 day
  Evaluation of hormone replacement therapy with glucocorticoids by a clinical score. Hypothesis: Patients with chronic adrenal insufficiency and a high frequency of adrenal crisis suffer from under-replacement.
Replacement therapy with mineralocorticoids | 1 day
  Evaluation of hormone replacement therapy with mineralocorticoids by a clinical and biochemical assessment. Hypothesis: Patients with chronic adrenal insufficiency and a high frequency of adrenal crisis suffer from under-replacement.
Glucocorticoid-receptor-polymorphisms | 1 day
  Evaluation of glucocorticoid-receptor-polymorphisms (ER 22/23 EK, N363S, bcl1, 9beta, Tth3l). Hypothesis: Patients with chronic adrenal insufficiency and a high frequency of adrenal crisis have a higher prevalence of glucocorticoid-receptor-polymorphisms.
Catecholamine-levels | 1 day
  Evaluation of catecholamine-levels (ng/l). Hypothesis: Patients with chronic adrenal insufficiency and a high frequency of adrenal crisis have a more pronounced catecholamin-deficit.
Patient education | 1 day
  Evaluation of patient education by questionnaire. Hypothesis: Patients with chronic adrenal insufficiency and a high frequency of adrenal crisis have a worse education status.

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Hahner, MD, Prof., Principal Investigator — Univesity Hospital Wuerzburg
Locations (1):
- University Hospital Wuerzburg, Dept. of medicine I, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hahner S, Spinnler C, Fassnacht M, Burger-Stritt S, Lang K, Milovanovic D, Beuschlein F, Willenberg HS, Quinkler M, Allolio B. High incidence of adrenal crisis in educated patients with chronic adrenal insufficiency: a prospective study. J Clin Endocrinol Metab. 2015 Feb;100(2):407-16. doi: 10.1210/jc.2014-3191. Epub 2014 Nov 24. PMID 25419882
- [Background] Allolio B. Extensive expertise in endocrinology. Adrenal crisis. Eur J Endocrinol. 2015 Mar;172(3):R115-24. doi: 10.1530/EJE-14-0824. Epub 2014 Oct 6. PMID 25288693
- [Background] Reisch N, Willige M, Kohn D, Schwarz HP, Allolio B, Reincke M, Quinkler M, Hahner S, Beuschlein F. Frequency and causes of adrenal crises over lifetime in patients with 21-hydroxylase deficiency. Eur J Endocrinol. 2012 Jul;167(1):35-42. doi: 10.1530/EJE-12-0161. Epub 2012 Apr 18. PMID 22513882
- [Background] Reincke M, Ritzel K, Osswald A, Berr C, Stalla G, Hallfeldt K, Reisch N, Schopohl J, Beuschlein F. A critical reappraisal of bilateral adrenalectomy for ACTH-dependent Cushing's syndrome. Eur J Endocrinol. 2015 Oct;173(4):M23-32. doi: 10.1530/EJE-15-0265. Epub 2015 May 20. PMID 25994948
- [Background] Smans LC, Van der Valk ES, Hermus AR, Zelissen PM. Incidence of adrenal crisis in patients with adrenal insufficiency. Clin Endocrinol (Oxf). 2016 Jan;84(1):17-22. doi: 10.1111/cen.12865. Epub 2015 Aug 27. PMID 26208266
- [Background] Hahner S, Arlt W, Allolio B. [Adrenal crisis. Diagnostic and therapeutic management of acute adrenal cortex insufficiency]. Internist (Berl). 2003 Oct;44(10):1243-52. doi: 10.1007/s00108-003-1050-1. German. PMID 14689086